CLINICAL TRIAL: NCT02761967
Title: Physical Training in Water (SWEP Method) During Pregnancy and Low Pressure Fitness (LPF) in Postpartum Period, Effects on Women
Brief Title: Physical Activity in Pregnancy and Postpartum Period, Effects on Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Carlos Sanchez Garcia (Other)
Responsible Party: Sponsor-Investigator, Juan Carlos Sanchez Garcia, PhD, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20022014UGR
Record Dates: First submitted 2016-04-25; First posted 2016-05-04 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Pregnancy
Keywords: Physical activity; Pregnancy; Childbirth; Postpartum period; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity (Experimental): The women in the EG (Exercise Group) performed moderate physical exercise in water, following the SWEP method (Study of Water-based Exercise during Pregnancy). It consists of performing moderate physical exercise in an aquatic environment from weeks 20 to 37 of gestation. The sessions take place three times weekly, with a duration of 60 minutes each (45 minutes of activity followed by 15 minutes of relaxation). The sessions are composed of three phases: a) warm-up; b) the main phase, divided into aerobic exercise and strength-endurance exercises, designed specifically for pregnant women; c) stretching and relaxation.
  After the postpartum period, women begin a program based on postpartum recovery exercises Fitness Low Pressure method 12-week, 3 days a week, in sessions of 60 minutes.
  Interventions: Behavioral: Physical activity
- No exercise (No Intervention): The CG (Control Group) received the standard recommendations during pregnancy, including guidelines from the midwife on the positive effects of physical exercise. These participants received the usual visits from healthcare providers (midwives, obstetricians and family doctor) during pregnancy, as did those in the EG.
  After the postpartum period, the women in the control group did not perform regulated physical activity.

INTERVENTIONS:
Behavioral: Physical activity — Women from the 20th week of moderate physical exercise performed in water character designed following the guidelines in the SWEP method will end in week 37 of gestation. After the postpartum period, women begin a program based on postpartum recovery exercises Fitness Low Pressure method 12-week, 3 days a week, in sessions of 60 minutes.
  Arms: Physical activity

SUMMARY:
This study evaluates whether the use of moderate physical exercise character in water is beneficial for pregnant women. Half of the participants will carry out moderate physical exercise character in water, following the protocol developed specifically for this purpose and called SWEP (Study Water Exercises Program) method, while the other group will not perform physical exercise during pregnancy.

Concluded the postpartum period, women perform exercises aimed postpartum recovery. The women's group has conducted exercises during pregnancy postpartum recovery made under the guidance of LPF (Low Pressure Fitness) method.

DETAILED DESCRIPTION:
Preliminary phase:

Current status of the subject.

During this phase will be an updated systematic search research topic. The literature search in databases such as MEDLINE, SCOPUS, CINAHL, WoS (Web Of Science) among others.

Data Collection: The source for the collection of primary data is through a personal interview with the participants and through the primer health of pregnant and/or medical history.

Interview on the first visit:

* Collect socioeconomic and health data about participants: age, parity, weight, BMI, smoking habits, drug use, profession/occupation, education level, physical activity pattern prior to pregnancy.
* Degree of overall health perception.
* Assess the risks according to the guide of the American College of Obstetricians and Gynecologists.
* Obtaining informed when agreeing to participate in the study consent.
* Give information pack about the exercises that the investigators will perform well as controls to be made in each session, and general rules to practice any physical activity.

Execution:

Classes are held in the morning hours preferable between 10 and 11 o'clock in the morning after a caloric intake and adequate hydration.

Every participant should carry your water bottle during each session that will take place, as well as adequate clothing, in which bathing suit, hat, glasses and proper footwear is included to prevent falls.

Before each class dynamics to follow and the signs that will make the exercise should stop, every participant should know how to take her own pulse at the level of the carotid artery may recall, because at different times of the central activity will take frequency heart, as a general rule must be able to hold a conversation without much difficulty while performing the exercise, and during the performance of this should properly hydrated according to the needs of each one in particular.

1. Warm up: The warm-up exercise will take place in a small vessel, where the water depth is around the thighs.

   The session starts with the upper body and decreasing order to heat the lower body.
2. Central part of the activity. It is be held in the large vessel, exercise intensity will increase in order to keep within the limits for an exercise of moderate, use different devices support to carry it out and exercises of strength, endurance and pelvic elasticity are included.

   Assistive devices that will use floating elements that will help us reduce the intensity of exercise providing flotation and will serve as support material to work specific parts. These devices are floating tables expanded polystyrene foam boys pull soft polyethylene and flexible floating bars and playful elements, such as balls, rings, ... spades.
3. Phase cool down. In this phase the participants will seek to return to calm, will be done in the small vessel having 3-4 ° C more than the large glass. exercises to progressively reducing the intensity and ending with relaxation exercises will be conducted .

The exercises are flexibility the investigators will not keep avoiding positions that strain the joints due to the state of gestation, those areas that have been previously exercised not to exceed the natural movement will stretch.

Once found befallen birth one review and extraction of data on birth process will take place and will take a final interview with the participant to collect data that will be obtained during the postpartum period such as type of feed received by the newborn, and value the existence of postpartum depression with the Edinburgh test.

Concluded the postpartum period. Women begin a program of recovery postpartum 12 weeks, 3 times a week in sessions of one hour. They perform warm-up exercises, a central part of Low Pressure Fitness exercises and end with stretching exercises.

ELIGIBILITY:
Inclusion Criteria:

* Do not suffer any absolute contraindications according to the American College of Obstetricians and Gynecologists.
* If there is a relative contraindication, participation in the intervention group should be favorable report by participants obstetrician.
* To know how to swim.
* To sign informed consent to participate in research consent.

Exclusion Criteria:

* Absolute contraindications to aerobic exercise during pregnancy.

  * Restrictive lung disease.
  * Heart disease with hemodynamic consequences.
  * Incompetent cervix/cerclage.
  * Multiple gestation with preterm labor.
  * Persistent bleeding in the second or third trimester bleeding.
  * Previa after 26 weeks of gestation.
  * Preterm birth during the current pregnancy.
  * Rupture of membranes.
  * Pregnancy-induced hypertension.
* Relative contraindications to aerobic exercise during pregnancy.

  * Severe anemia.
  * Cardiac arrhythmia maternal unevaluated.
  * Chronic Bronchitis.
  * Type I diabetes poorly controlled.
  * Extreme morbid obesity.
  * Under extreme weight (BMI <12).
  * History of extremely sedentary life style.
  * Intrauterine growth restriction in current pregnancy.
  * Poorly controlled hypertension / pre-eclampsia.
  * Orthopedic limitations.
  * Poorly controlled seizure disorders.
  * Poorly controlled Thyroid disease.
  * Heavy smoker.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2016-11-12 (Actual); Study Completion 2017-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MARIA JOSE AGUILAR CORDERO, Principal Investigator — UNIVERSITY OF GRANADA (SPAIN)
Locations (1):
- Instituto Mixto Universitario Deporte y Salud, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aguilar-Cordero MJ, Sanchez-Garcia JC, Rodriguez-Blanque R, Sanchez-Lopez AM, Mur-Villar N. Moderate Physical Activity in an Aquatic Environment During Pregnancy (SWEP Study) and Its Influence in Preventing Postpartum Depression. J Am Psychiatr Nurses Assoc. 2019 Mar/Apr;25(2):112-121. doi: 10.1177/1078390317753675. Epub 2018 Feb 28. PMID 29490560

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Activity: 1. º Phase: Swep Method. Warm up: The warm-up exercise will take place in a small vessel, where the water depth is around the thighs.
     Central part of the activity: It is be held in the large vessel, exercise intensity will increase in order to keep within the limits for an exercise of moderate, use different devices support to carry it out and exercises of strength, endurance and pelvic elasticity are included.
     Phase cool down: In this phase the participants will seek to return to calm, will be done in the small vessel having 3-4 ° C more than the large glass. exercises to progressively reducing the intensity and ending with relaxation exercises will be conducted .
  2. º Phase: Low Pressure Fitness. Concluded the postpartum period. Women begin a program of recovery postpartum 12 weeks, 3 times a week in sessions of one hour. They perform warm-up exercises, a central part of Low Pressure Fitness exercises and end with stretching exercises.
- No Exercise: Not take place during the gestation period between gestation week 20 to 37 any physical exercise.
  Not take place during the postpartum period any physical exercise.
Period: Overall Study
Arm/Group | Physical Activity | No Exercise
Started | 70 | 70
Completed | 65 | 64
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Physical Activity: The woman he joins the intervention group meets once a week 20 of gestation and ends after serving 37 weeks. Intervention will consist of physical exercise of moderate character in water, according to the methodology of the method of SWEP, for an hour a day, three days a week.
  After the postpartum period, women begin a program based on postpartum recovery exercises Fitness Low Pressure method 12-week, 3 days a week, in sessions of 60 minutes.
  Physical activity: Women from the 20th week of moderate physical exercise performed in water character designed following the guidelines in the SWEP method will end in week 37 of gestation. After the postpartum period, women begin a program based on postpartum recovery exercises Fitness Low Pressure method 12-week, 3 days a week, in sessions of 60 minutes.
- Total: Total of all reporting groups
Arm/Group | Physical Activity | No Exercise | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 70 | 140
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.74 (4.41) | 33.47 (5.18) | 34.1 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 140
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 70 | 70 | 140
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.7 (4.16) | 24.93 (4.80) | 24.81 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Delivery Times Measured in Partogram
Description: This result is to measure the difference in time between births to women who have made physical exercise during pregnancy, SWEP method, compared to women who have not exercised .
Time Frame: Twenty four month
Population: The total duration of delivery times between women in the control group and women in the exercise group will be compared.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Physical Activity: The women in the EG performed moderate physical exercise in water, following the SWEP method (Study of Water-based Exercise during Pregnancy). It consists of performing moderate physical exercise in an aquatic environment from weeks 20 to 37 of gestation. The sessions take place three times weekly, with a duration of 60 minutes each (45 minutes of activity followed by 15 minutes of relaxation). The sessions are composed of three phases: a) warm-up; b) the main phase, divided into aerobic exercise and strength-endurance exercises, designed specifically for pregnant women; c) stretching and relaxation.
  After the postpartum period, women begin a program based on postpartum recovery exercises Fitness Low Pressure method 12-week, 3 days a week, in sessions of 60 minutes.
- No Exercise: The CG received the standard recommendations during pregnancy, including guidelines from the midwife on the positive effects of physical exercise. These participants received the usual visits from healthcare providers (midwives, obstetricians and family doctor) during pregnancy, as did those in the EG.
  After the postpartum period, the women in the control group did not perform regulated physical activity.
Arm/Group | Physical Activity | No Exercise
Number analyzed (Participants) | 60 | 60
minutes | 389.33 (216.18) | 561.3 (199.94)
Statistical Analysis 1: Comparison: Physical Activity vs No Exercise; Test type: Equivalence — The statistical power of the study for the temporal variables was 82%. Multiple linear regression models were obtained for the first and second stages and for the total duration of delivery; p = 0.776, Chi-squared

2. Primary Outcome: Edinburgh Postnatal Depression Scale
Description: Determine the rate of postpartum depression in both groups. The scale consists of ten short questions, all of which must be answered. The subject is asked to choose, of the four possible answers, the one that most closely describes how she felt during the week prior to the test. The response options range from 0 (for example, no, not at all or no, never again) to 3 (for example, yes, most of the time or yes, very often). The total score is recorded in a table ranging from 0 to 30, where higher values indicate more severe symptoms of depression.
  For this study, total scores below 10 were classed as "no risk" and scores of 10 or more indicated the presence of risk. Scores above 16 indicated a more severe risk of depression, and suggested that additional evaluations should be conducted immediately.
Time Frame: Six month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Physical Activity: The woman he joins the intervention group meets once a week 20 of gestation and ends after serving 37 weeks. Intervention will consist of physical exercise of moderate character in water, according to the methodology of the SWEP method, for an hour a day, three days a week.
  After the postpartum period, women begin a program based on postpartum recovery exercises Fitness Low Pressure method 12-week, 3 days a week, in sessions of 60 minutes.
  Physical activity: Women from the 20th week of moderate physical exercise performed in water character designed following the guidelines in the SWEP method will end in week 37 of gestation. After the postpartum period, women begin a program based on postpartum recovery exercises Fitness Low Pressure method 12-week, 3 days a week, in sessions of 60 minutes.
Arm/Group | Physical Activity | No Exercise
Number analyzed (Participants) | 70 | 70
units on a scale | 6 (3.39) | 8 (2.33)

3. Secondary Outcome: Sleep Quality in Pregnant; Pittsburgh Sleep Quality Index (PSQI)
Description: Assess the quality of sleep of pregnant women with moderate activity in water, with respect to who do not practice.
  Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.The order of the PSQI items has been modified from the original order in order to fit the first 9 items (which are the only items that contribute to the total score) on a single page. Item 10, which is the second page of the scale, does not contribute to the PSQI score.
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: Twelve month
Population: During the data collection, 3 women from the control group were lost because they did not complete the PSQI questionnaire during the follow-up phase. The analysis excluded 3 women from the intervention group due to errors at the time of completing the PSQI questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity | No Exercise
Number analyzed (Participants) | 67 | 67
units on a scale | 6.84 (2.86) | 10.10 (3.12)

ADVERSE EVENTS:
Arm/Group | Physical Activity | No Exercise
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No